CLINICAL TRIAL: NCT05211024
Title: A Follow-up Study for Patients Who Participated in the GOAL Trial (GOAL-Post)
Brief Title: A Long-term Follow up Study for Patients Who Participated in the GOAL Trial (GOAL-Post)
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Uganda Heart Institute (Other); Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0451
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Rheumatic Heart Disease
MeSH Terms: conditions — Rheumatic Heart Disease | interventions — Penicillin G Benzathine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, RNA, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aim 1: Group A: Children and adolescent who are prior GOAL participants who have a normal echocardiogram at the 2 year endpoint and are no receiving secondary antibiotic prophylaxis
- Aim 1 Group B: Children and adolescent who have a normal echocardiogram at the start of the study
- Aim 2: Children and adolescent who are prior GOAL participants who have persistent latent RHD on echocardiogram at the 2 year endpoint.
  Interventions: Drug: Penicillin G Benzathine

INTERVENTIONS:
Drug: Penicillin G Benzathine — Participants in Aim 2 are receiving 28 days interval BPG intramuscular injection as part of standard of care
  Groups: Aim 2

SUMMARY:
GOAL-Post is comprised of two studies that will help refine recommendations for the duration of secondary prophylaxis for children diagnosed with latent RHD, which is currently not known

DETAILED DESCRIPTION:
GOAL-Post is comprised of two studies that will help refine recommendations for the duration of secondary prophylaxis for children diagnosed with latent RHD, which is currently not known.

Aim 1: Compare the two-year risk of developing RHD (borderline or definite) between children and adolescents who completed the GOAL Trial with a normal echocardiogram (prior diagnosis of latent RHD) and age/sex/and geographically matched controls with repeated normal echocardiograms (normal in both the original GOAL screening in 2017/2018 and in the planned GOAL-Post screening in 2021).

Aim 2: Determine the five-year rate of RHD progression and regression among children with persistent latent RHD who receive secondary antibiotic prophylaxis (medium-term impact of prophylaxis). Five years includes time from initial GOAL enrollment to the end of GOAL-Post.

Aim 3: Create a RHD biobank that will support further research on RHD genetic susceptibility and pathophysiology

ELIGIBILITY:
Inclusion Criteria:

Aim 1: Group A: Children and adolescents will be eligible for Aim 1 if they (1) are a prior GOAL participant deemed by the adjudication panel to have a normal echocardiogram at the 2-year endpoint, (2) are not receiving secondary antibiotic prophylaxis, and (3) agree to participate in the study via the study's informed consent/assent process.

Group B: Children and adolescents will be eligible for Aim 1 if they (1) have a normal echocardiogram at the start of the study, (2) Meet the age/sex/geographic match requirement (from former GOAL participants), and (3) have agreed to participate in the study via the study's informed consent/assent process.

Aim 2: Children and adolescents will be eligible for Aim 2 if they (1) are a prior GOAL participant deemed by the adjudication panel to have persistent latent RHD on echocardiogram at the 2-year endpoint, (2) have been prescribed secondary antibiotic prophylaxis, and (3) agree to participate in the study via the study's informed consent/assent process.

Aim 3: Children and adolescents will be eligible for Aim 3 if they are prior GOAL participants deemed by the adjudication panel to (1) have a normal echocardiogram at the 2-year endpoint (Aim 1 participants), (2) deemed by the adjudication panel to have persistent latent RHD at the 2-year endpoint (Aim 2 participants), or (3) deemed by the adjudication panel to have moderate/severe RHD at the 2-year endpoint. Aim 3 will include a separate consent/assent and participants will be able to participate in each aim independently.

Exclusion Criteria:

Aim 1: Group A: Residence or school is no longer in Gulu District or one of the surrounding districts.

Group B: Known history of ARF or RHD, or evidence of RHD on baseline echocardiogram or structural or functional cardiac defects, other than those consistent with RHD, that were known prior to or detected through echo screening (except patent foramen ovale, small atrial septal defect, small ventricular septal defect, small patent ductus arteriosus).

Aim 2 + 3: Residence or school is no longer in Gulu District or one of the surrounding districts.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Aim 1 will enroll with normal echocardiograms after 2-years of participation in the GOAL Trial (Group A) and an appropriate number of age/sex matched controls (Group B) without echocardiographic evidence of RHD.
  Aim 2 will enroll participants with persistent latent RHD after 2 years of participation in the GOAL Trial. (Fig. 2).
Sampling Method: Probability Sample
Enrollment: 1423 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Progression | 2 year endpoint
  Progression of echocardiographic features of latent RHD to borderline to definite, or definite to mild or definitive to moderate/severe
Regression | 2 year endpoint
  Regression of echocardiographic features of latent RHD

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Z Beaton, MD, Principal Investigator — Cincinnati Chidren's hospital
Locations (1):
- Uganda Heart Institute, Kampala, Uganda

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-07-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT05211024/SAP_000.pdf